CLINICAL TRIAL: NCT00988338
Title: A Radiographic and Clinical Study Evaluating a Novel Allogeneic, Cancellous, Bone Matrix Containing Viable Stem Cells (Trinity Evolution Matrix) in Subjects Undergoing Foot and Ankle Fusion
Brief Title: Evaluation of Trinity Evolution in Patients Undergoing Foot and Ankle Fusion
Acronym: TAF
Status: Completed | Type: Observational
Sponsor: Orthofix Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TY01AF
Record Dates: First submitted 2009-09-29; First posted 2009-10-02 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Tibiotalar Arthrodesis; Subtalar Arthrodesis; Calcaneocuboid Arthrodesis; Talonavicular Arthrodesis; Double Arthrodesis (i.e. Calcaneocuboid and Talonavicular); Triple Arthrodesis (i.e. Subtalar, Calcaneocuboid, and Talonavicular)
Keywords: Trinity Evolution; Arthrodesis; Foot Fusion; Ankle Fusion; Allograft
MeSH Terms: conditions — Ankylosis | interventions — Transplantation, Homologous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Trinity Evolution
  Interventions: Biological: Trinity Evolution

INTERVENTIONS:
Biological: Trinity Evolution — Novel Allogeneic, Cancellous, Bone Matrix Containing Viable Stem and Osteoprogenitor Cells
  Other Names: Allograft; Mesenchymal Stem Cells

SUMMARY:
The purpose of this study is to utilize Trinity Evolution as a graft source in foot/ankle fusions and to follow the subjects to measure the clinical outcomes and fusion rate. The hypothesis of the study is that Trinity Evolution will result in fusion rates and clinical outcomes similar to those obtained from autograft and other routinely used allograft materials; these include: fusion, improvement in pain, improvement in function, and absence of adverse events related to the use of the graft source.

DETAILED DESCRIPTION:
Symptomatic arthritic conditions of the foot and ankle including osteoarthritis, post-traumatic arthritis, inflammatory arthropathies and others can be painful and disabling conditions that lead to a reduced quality of life. Major symptoms include pain, stiffness, swelling, and difficulty walking. Many patients may be initially treatable with non-invasive measures such as analgesics, ankle-foot orthosis, physical therapy and medications such as steroids; however, over time, surgery becomes necessary to improve quality of life and maintain function. Arthrodesis is a well-known procedure that can reduce pain and result in a foot/ankle that can withstand an active lifestyle.

Bone graft is used to stimulate new bone formation at the operative site by providing osteogenic cells with osteoinductive factors with an osteoconductive matrix. Although autologous bone is often used as the structural graft material for fusion procedures, donor site morbidity (e.g., pain, infection, and fracture), limited supply, and inconsistent osteogenic activity continue to be associated problems. The quality of an autograft is dependent upon the age and medical condition of the patient, as well as the number of viable mesenchymal and osteoprogenitor stem cells that are present in the specimen. This tissue is harvested during the surgical procedure; the process can prolong morbidity at the harvest site. The ideal bone graft would offer osteogenic cells, osteoinductive factors, and an osteoconductive matrix with a consistent supply of viable mesenchymal stem cells (MSCs) and osteoprogenitor cells (OPCs)-but without the morbidity of autograft.

Due to the limitations associated with autograft, researchers are pursuing the use of bone-graft substitutes to promote arthrodesis. Bone-graft substitutes now being used by surgeons include ceramic synthetics, bone morphogenic proteins (BMPs), demineralized bone matrices (DBMs) and other allografts; these may be used alone or in combination. Allografts available as substitutes for autograft offer some of the benefits of autograft without its limitations-but do not contain viable MSCs and OPCs.

Trinity Evolution is an allogeneic cancellous bone matrix containing demineralized cortical bone (DCB) as well as viable osteoprogenitor and mesenchymal stem cells. Adult mesenchymal stem cells and osteoprogenitor cells, such as those in Trinity Evolution, are the precursor cells that differentiate into osteoblasts-the cells responsible for bone growth and repair.

Trinity Evolution provides the required osteoconduction, osteogenesis, and osteoinductivity necessary for successful bone grafting. It offers viable osteoprogenitor and mesenchymal stem cells and demineralized cortical bone-all in a single product. Data from preclinical studies with Trinity Evolution have demonstrated in-vitro and in-vivo safety and effectiveness. Trinity Evolution is a "minimally manipulated" tissue that is considered an allograft, and as such, is labeled for bone repair for all orthopedic and podiatric indications where autograft is used. In this study, Trinity Evolution will be used as a substitute for autograft and/or standard allograft in the following arthrodesis procedures: tibiotalar, subtalar, calcaneocuboid, talonavicular, double fusions (i.e. calcaneocuboid and talonavicular), and triple fusions (i.e. subtalar, calcaneocuboid, and talonavicular).

ELIGIBILITY:
Inclusion Criteria:

* Foot and/or ankle pathology requiring fusion using open surgical technique with supplemental bone graft/substitute requiring one of the following procedures:

  * Ankle joint fusion
  * Subtalar fusion
  * Calcaneocuboid fusion
  * Talonavicular fusion
  * Double fusions (talonavicular and calcaneocuboid joints)
  * Triple fusions (subtalar, talonavicular, and calcaneocuboid joints)
* At least 18 years of age
* Willing and able to comply with the requirements of the protocol including follow-up requirements
* Willing and able to sign a study-specific informed consent.

Exclusion Criteria:

* Use of any other bone graft or bone graft substitute in addition to or in place of Trinity Evolution at the time of surgery
* Use of adjunctive post-operative stimulation
* Active local or systemic infection
* Currently pregnant or considering becoming pregnant during the follow-up period
* Active malignancy or having been on chemotherapy of any kind for a malignancy in the past 1 year
* Immunosuppressive therapy of any kind within the past 1 year
* Has a known history of hypersensitivity or anaphylactic reaction to dimethyl sulfoxide (DMSO).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject selection will be determined by orthopedic surgeon.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2009-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Fusion Success | 12 months

SECONDARY OUTCOMES:
Improvement in scores: Ankle-Hindfoot Scale (AHS), Visual Analog Scale (VAS), and Health Survey (SF-36v2). | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Raymond J Linovitz, MD, Study Director — Orthofix Inc.
Locations (10):
- United States (10):
  - Orthopaedic Associates of South Broward, PA, Hollywood, Florida
  - Sinai Hospital of Baltimore / Rubin Institute for Advanced Orthopedics, Baltimore, Maryland
  - New Mexico Orthopedics, Albuquerque, New Mexico
  - OrthoCarolina Research Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Ohio Orthopedic Center of Excellence, Upper Arlington, Ohio
  - The Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - Central Tennessee Foot and Ankle Center, Sparta, Tennessee
  - Franciscan Foot and Ankle Specialists, Burien, Washington